CLINICAL TRIAL: NCT05064384
Title: Axonics SacRal NeuromodulaTIon System RegisTRY Study : ARTISTRY
Brief Title: Axonics SacRal NeuromodulaTIon System RegisTRY Study
Acronym: ARTISTRY
Status: Completed | Type: Observational
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 105-0076
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Urinary Retention; Urinary Urge Incontinence; Urgency-Frequency; Fecal Incontinence
Keywords: Overactive Bladder, bladder control, bowel control
MeSH Terms: conditions — Urinary Retention; Urinary Incontinence, Urge; Fecal Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
To assess the post-market clinical outcomes with use of the Axonics Sacral Neuromodulation System(s).

DETAILED DESCRIPTION:
The study will be a prospective, multi-center, single-arm, post-market registry study. Participant outcomes will be compared to their baseline, with participants serving as their own control.

The study is expected to complete enrollment in approximately 24 months and follow the patients per protocol for 1 year. The study was conducted at approximately 30 centers in the United States and Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to be trialed with the Axonics External Trial System (ETS), or patients scheduled to receive an Axonics Implantable neurostimulator (INS) or Axonics FS implant
2. Willing and capable of providing informed consent
3. Capable of participating in all testing associated with this clinical investigation

Exclusion Criteria:

For all indications:

1. Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound evaluation of study endpoints
2. Any psychiatric or personality disorder at the discretion of the study physician
3. History of allergic response to titanium, zirconia, polyurethane, epoxy, or silicone
4. A female who is breastfeeding
5. A female with a positive urine pregnancy test

   For OAB & UR:
6. Current urinary tract mechanical obstruction (e.g. benign prostatic enlargement or urethral stricture)
7. Current symptomatic urinary tract infection (UTI)

   For FI only:
8. Rectomucosal prolapse or congenital anorectal malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are scheduled to undergo an Axonics Trial or Axonics System will be considered candidates for the study and will be recruited from each Investigator's patient population.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Study Director — Axonics, Inc.
Locations (27):
- United States (26):
  - Arkansas Urology Research Center, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - Stanford Medicine, Redwood City, California
  - Sansum Clinic Urology, Santa Barbara, California
  - Manatee Medical Research Institute, Bradenton, Florida
  - Urologic Solutions, Fort Myers, Florida
  - Florida Urology Partners, North Redington Beach, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - Florida Urology Partners, Tampa, Florida
  - Northwestern, Chicago, Illinois
  - LSU Health, New Orleans, Louisiana
  - Ochsner Health, New Orleans, Louisiana
  - Chesapeake Urology, Hanover, Maryland
  - Comprehensive Urology, Royal Oak, Michigan
  - Adult Pediatric Urology & Urogynecology, Omaha, Nebraska
  - The Urology Center PC, Omaha, Nebraska
  - New Jersey Urology, Englewood, New Jersey
  - Stony Brook University, Stony Brook, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Urologic Specialists Oklahoma, Tulsa, Oklahoma
  - Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Penn State University, Hershey, Pennsylvania
  - The Female Pelvic Health Center, Newtown, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Southern Urogynecology, West Columbia, South Carolina
  - Center for Pelvic Health, Franklin, Tennessee
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-randomized study recruited participants who may have had an overlap of their diagnoses, some of which the overlap could have been as a result of their responses to certain questionnaires. For example, participants who scored ≥6 on the CCF-FIS questionnaires at baseline would be included in the FI cohort analysis while their primary indication may be UUI. Because of this, the numbers in the Participant Flow are not able to be stratified into each type of diagnosis.
Groups:
- Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI): Patients diagnosed with overactive bladder (OAB), urinary retention (UR), and/or fecal incontinence (FI) who underwent an Axonics External Trial System (ETS) trial surgery and/or full system implant surgery of the Axonics Implantable Neurostimulator (INS).
Period: Screening
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
Started | 272
Completed | 268
Not Completed | 4
Period: Safety
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
Started | 268
Completed | 253
Not Completed | 15
Period: Treatment
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
Started | 253
Completed | 250
Not Completed | 3
Period: Implant
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
Started | 250
Completed | 218
Not Completed | 32

BASELINE CHARACTERISTICS:
Population: Characteristics of the Treated study population. Participants in the Treated analysis population are those who were implanted with PNE or tined leads.
Groups:
- Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI): Patients diagnosed with overactive bladder (OAB), urinary retention (UR), and/or fecal incontinence (FI) who were scheduled to undergo an Axonics External Trial System (ETS) trial or receive an Axonics Implantable Neurostimulator (INS).
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 153
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 240
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 23
  Race: American Indian or Alaska Native | 1
  Race: Asian | 2
  Race: Caucasian | 217
  Race: Latino or Hispanic | 5
  Race: Other | 1
  Race: Declined to state | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 250
BMI [Number; unit: participants]
  < 18.5 kg/m2 | 2
  18.5-24.9 kg/m2 | 42
  25.0-29.9 kg/m2 | 79
  30.0-34.9 kg/m2 | 60
  35.0-39.9 kg/m2 | 28
  >=40.0 kg/m2 | 25
  Unknown | 14

OUTCOME MEASURES:

1. Primary Outcome: Therapy Responder Rate
Description: Percentage of participants who were determined as responders by the treating physician when using the External Trial Stimulator and who received the Axonics System. At least a 50% reduction in symptoms is considered standard in relevant literature for response rate therefore decision for determination of responder was left to PI discretion.
Time Frame: External Trial System Evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
Number analyzed (Participants) | 218
Participants | 206

2. Primary Outcome: Performance/Effectiveness - Improvement of Patient UUI Symptoms in the Implanted Cohort From Baseline
Description: Change in indication-specific patient symptoms from baseline for all implanted patients by Patient Symptom Questionnaire results. The patient symptoms questionnaire assesses participants' diagnosis-specific symptoms at baseline and at follow-up. Participants who reported a UUI diagnosis at baseline were asked about the number of urgency leaks experienced.
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: leaks per day
Groups:
- Overactive Bladder (OAB) - Urinary Urge Incontinence (UUI): Patients diagnosed with overactive bladder (OAB) who underwent an Axonics External Trial System (ETS) trial and received an Axonics Implantable Neurostimulator (INS) who experienced fewer leaks with less urgency.
Arm/Group | Overactive Bladder (OAB) - Urinary Urge Incontinence (UUI)
Number analyzed (Participants) | 182
leaks per day
  Baseline: Urgency leaks per day | 4.8 (6.1)
  6-month: Urgency leaks per day: number analyzed (Participants) | 152
  6-month: Urgency leaks per day | 2.4 (2.7)
  1-year: Urgency leaks per day: number analyzed (Participants) | 132
  1-year: Urgency leaks per day | 2.4 (3.6)

3. Primary Outcome: Performance/Effectiveness - Improvement of Patient UUI Symptoms in the Implanted Cohort From Baseline
Description: as for outcome 2
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: leaks after bed
Arm/Group | Overactive Bladder (OAB) - Urinary Urge Incontinence (UUI)
Number analyzed (Participants) | 182
leaks after bed
  Baseline: Urgency leaks after bed | 2.2 (2.8)
  6-month: Urgency leaks after bed: number analyzed (Participants) | 152
  6-month: Urgency leaks after bed | 1.1 (2.0)
  1-year: Urgency leaks after bed: number analyzed (Participants) | 132
  1-year: Urgency leaks after bed | 1.0 (2.0)

4. Primary Outcome: Performance/Effectiveness - Improvement of Patient UF Symptoms in the Implanted Cohort From Baseline
Description: Change in indication-specific patient symptoms from baseline for all implanted patients by Patient Symptom Questionnaire results. The patient symptoms questionnaire assesses participants' diagnosis-specific symptoms at baseline and at follow-up. Participants who reported a UF diagnosis at baseline were asked about the number of urinations they experienced per day and at night.
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: urinations per day
Groups:
- Overactive Bladder (OAB) - Urinary Frequency (UF): Patients diagnosed with overactive bladder (OAB) who underwent an Axonics External Trial System (ETS) trial and received an Axonics Implantable Neurostimulator (INS) who experienced fewer leaks with less urgency.
Arm/Group | Overactive Bladder (OAB) - Urinary Frequency (UF)
Number analyzed (Participants) | 151
urinations per day
  Baseline: Urinations per day | 8.8 (4.5)
  6-month: Urinations per day: number analyzed (Participants) | 125
  6-month: Urinations per day | 7.8 (8.0)
  1-year: Urinations per day: number analyzed (Participants) | 116
  1-year: Urinations per day | 6.7 (2.7)

5. Primary Outcome: Performance/Effectiveness - Improvement of Patient UF Symptoms in the Implanted Cohort From Baseline
Description: as for outcome 4
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: urinations at night
Arm/Group | Overactive Bladder (OAB) - Urinary Frequency (UF)
Number analyzed (Participants) | 151
urinations at night
  Baseline: Urinations at night | 3.0 (2.4)
  6-month: Urinations at night: number analyzed (Participants) | 125
  6-month: Urinations at night | 1.9 (2.2)
  1-year: Urinations at night: number analyzed (Participants) | 116
  1-year: Urinations at night | 2.0 (2.3)

6. Primary Outcome: Performance/Effectiveness - Improvement of Patient Urgency Symptoms in the Implanted Cohort From Baseline
Description: Change in indication-specific patient symptoms from baseline for all implanted patients by Patient Symptom Questionnaire results. The patient symptoms questionnaire assesses participants' diagnosis-specific symptoms at baseline and at follow-up. Participants who reported a UUI diagnosis at baseline were asked about the degree of urgency leaks experienced using the following scale: 0=no urgency; 1=mild urgency; 2= moderate urgency; 3=strong urgency and 4=severe urgency.
Time Frame: 6-months, 1-year
Population: Number of participants experiencing degree of urgency on a scale of 0-4, 0 meaning no urgency and 4 meaning severe urgency. Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Overactive Bladder (OAB) - Urinary Urge Incontinence (UUI)
Number analyzed (Participants) | 182
Participants
  Baseline: Average degree of urgency = 0 | 7
  Baseline: Average degree of urgency = 1 | 6
  Baseline: Average degree of urgency = 2 | 21
  Baseline: Average degree of urgency = 3 | 90
  Baseline: Average degree of urgency = 4 | 58
  6-month: Average degree of urgency = 0: number analyzed (Participants) | 152
  6-month: Average degree of urgency = 0 | 21
  6-month: Average degree of urgency = 1: number analyzed (Participants) | 152
  6-month: Average degree of urgency = 1 | 27
  6-month: Average degree of urgency = 2: number analyzed (Participants) | 152
  6-month: Average degree of urgency = 2 | 48
  6-month: Average degree of urgency = 3: number analyzed (Participants) | 152
  6-month: Average degree of urgency = 3 | 36
  6-month: Average degree of urgency = 4: number analyzed (Participants) | 152
  6-month: Average degree of urgency = 4 | 20
  1-year: Average degree of urgency = 0: number analyzed (Participants) | 132
  1-year: Average degree of urgency = 0 | 21
  1-year: Average degree of urgency = 1: number analyzed (Participants) | 132
  1-year: Average degree of urgency = 1 | 28
  1-year: Average degree of urgency = 2: number analyzed (Participants) | 132
  1-year: Average degree of urgency = 2 | 47
  1-year: Average degree of urgency = 3: number analyzed (Participants) | 132
  1-year: Average degree of urgency = 3 | 23
  1-year: Average degree of urgency = 4: number analyzed (Participants) | 132
  1-year: Average degree of urgency = 4 | 13

7. Primary Outcome: Performance/Effectiveness - Improvement of Patient Urinary Urgency Symptoms in the Implanted Cohort From Baseline
Description: Change in indication-specific patient symptoms from baseline for all implanted patients by Patient Symptom Questionnaire results. The patient symptoms questionnaire assesses participants' diagnosis-specific symptoms at baseline and at follow-up. Participants who reported a UF diagnosis at baseline were asked about the degree of urgency experienced using the following scale: 0=no urgency; 1=mild urgency; 2= moderate urgency; 3=strong urgency and 4=severe urgency.
Time Frame: 6-months, 1-year
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Overactive Bladder (OAB) - Urinary Frequency (UF)
Number analyzed (Participants) | 151
Participants
  Baseline: Average degree of urgency = 0 | 2
  Baseline: Average degree of urgency = 1 | 5
  Baseline: Average degree of urgency = 2 | 24
  Baseline: Average degree of urgency = 3 | 76
  Baseline: Average degree of urgency = 4 | 44
  6-month: Average degree of urgency = 0: number analyzed (Participants) | 125
  6-month: Average degree of urgency = 0 | 15
  6-month: Average degree of urgency = 1: number analyzed (Participants) | 125
  6-month: Average degree of urgency = 1 | 23
  6-month: Average degree of urgency = 2: number analyzed (Participants) | 125
  6-month: Average degree of urgency = 2 | 47
  6-month: Average degree of urgency = 3: number analyzed (Participants) | 125
  6-month: Average degree of urgency = 3 | 27
  6-month: Average degree of urgency = 4: number analyzed (Participants) | 125
  6-month: Average degree of urgency = 4 | 13
  1-year: Average degree of urgency = 0: number analyzed (Participants) | 116
  1-year: Average degree of urgency = 0 | 14
  1-year: Average degree of urgency = 1: number analyzed (Participants) | 116
  1-year: Average degree of urgency = 1 | 25
  1-year: Average degree of urgency = 2: number analyzed (Participants) | 116
  1-year: Average degree of urgency = 2 | 38
  1-year: Average degree of urgency = 3: number analyzed (Participants) | 116
  1-year: Average degree of urgency = 3 | 26
  1-year: Average degree of urgency = 4: number analyzed (Participants) | 116
  1-year: Average degree of urgency = 4 | 13

8. Primary Outcome: Performance/Effectiveness - Improvement of Patient FI Symptoms in the Implanted Cohort From Baseline
Description: Change in indication-specific patient symptoms from baseline for all implanted patients by Patient Symptom Questionnaire results. The patient symptoms questionnaire assesses participants' diagnosis-specific symptoms at baseline and at follow-up. Participants who reported a FI diagnosis at baseline were asked about the number of FI episodes experienced.
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: episodes per week
Groups:
- Fecal Incontinence (FI): Patients diagnosed with Fecal Incontinence (FI) who underwent an Axonics External Trial System (ETS) trial and received an Axonics Implantable Neurostimulator (INS) who experienced fewer leaks with less urgency.
Arm/Group | Fecal Incontinence (FI)
Number analyzed (Participants) | 54
episodes per week
  Baseline: FI episodes per week | 6.3 (8.6)
  6-month: FI episodes per week: number analyzed (Participants) | 44
  6-month: FI episodes per week | 1.5 (2.7)
  1-year: FI episodes per week: number analyzed (Participants) | 35
  1-year: FI episodes per week | 2.4 (4.1)

9. Primary Outcome: Performance/Effectiveness - Improvement of Patient FI Symptoms in the Implanted Cohort From Baseline
Description: as for outcome 8
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Fecal Incontinence (FI)
Number analyzed (Participants) | 54
days per week
  Baseline: FI days per week | 3.8 (2.2)
  6-month: FI days per week: number analyzed (Participants) | 44
  6-month: FI days per week | 1.1 (1.7)
  1-year: FI days per week: number analyzed (Participants) | 35
  1-year: FI days per week | 1.8 (2.3)

10. Primary Outcome: Performance/Effectiveness - Improvement of Patient FI Urgency Symptoms in the Implanted Cohort From Baseline
Description: Change in indication-specific patient symptoms from baseline for all implanted patients by Patient Symptom Questionnaire results. The patient symptoms questionnaire assesses participants' diagnosis-specific symptoms at baseline and at follow-up. Participants who reported a FI diagnosis at baseline were asked about the degree of urgency experienced.
Time Frame: 6-months, 1-year
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Fecal Incontinence (FI): Patients diagnosed with Fecal Incontinence (FI) who underwent an Axonics External Trial System (ETS) trial and received an Axonics Implantable Neurostimulator (INS) who experienced fewer FI episodes with less urgency.
Arm/Group | Fecal Incontinence (FI)
Number analyzed (Participants) | 54
Participants
  Baseline: Average degree of urgency = 0 | 9
  Baseline: Average degree of urgency = 1 | 1
  Baseline: Average degree of urgency = 2 | 10
  Baseline: Average degree of urgency = 3 | 17
  Baseline: Average degree of urgency = 4 | 17
  6-month: Average degree of urgency = 0: number analyzed (Participants) | 44
  6-month: Average degree of urgency = 0 | 15
  6-month: Average degree of urgency = 1: number analyzed (Participants) | 44
  6-month: Average degree of urgency = 1 | 7
  6-month: Average degree of urgency = 2: number analyzed (Participants) | 44
  6-month: Average degree of urgency = 2 | 7
  6-month: Average degree of urgency = 3: number analyzed (Participants) | 44
  6-month: Average degree of urgency = 3 | 10
  6-month: Average degree of urgency = 4: number analyzed (Participants) | 44
  6-month: Average degree of urgency = 4 | 5
  1-year: Average degree of urgency = 0: number analyzed (Participants) | 35
  1-year: Average degree of urgency = 0 | 13
  1-year: Average degree of urgency = 1: number analyzed (Participants) | 35
  1-year: Average degree of urgency = 1 | 5
  1-year: Average degree of urgency = 2: number analyzed (Participants) | 35
  1-year: Average degree of urgency = 2 | 8
  1-year: Average degree of urgency = 3: number analyzed (Participants) | 35
  1-year: Average degree of urgency = 3 | 3
  1-year: Average degree of urgency = 4: number analyzed (Participants) | 35
  1-year: Average degree of urgency = 4 | 6

11. Primary Outcome: Performance/Effectiveness - Improvement in Quality of Life Scoring for OAB Participants in the Implanted Cohort
Description: Change in ICIQ-OABqol scores at follow-up compared to baseline for implanted participants. Questions in each subscale are scored by a summed range of 0 to 100, with a higher score indicating better quality of life. Overall score ≥ 10 points from baseline to follow-up is considered a minimally important difference (MID).
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Overactive Bladder (OAB): Patients diagnosed with overactive bladder (OAB)who underwent an Axonics External Trial System (ETS) trial and received an Axonics Implantable Neurostimulator (INS) that had a higher score than baseline and had a score change of 10 points or greater.
Arm/Group | Overactive Bladder (OAB)
Number analyzed (Participants) | 199
score on a scale
  Baseline: Coping | 49.4 (27.7)
  Baseline: Concern | 49.2 (25.0)
  Baseline: Sleep | 53.4 (29.0)
  Baseline: Social | 75.0 (22.5)
  Baseline: HRQL | 55.3 (22.3)
  6-Month: Coping: number analyzed (Participants) | 168
  6-Month: Coping | 74.8 (26.2)
  6-Month: Concern: number analyzed (Participants) | 168
  6-Month: Concern | 74.8 (25.1)
  6-Month: Sleep: number analyzed (Participants) | 168
  6-Month: Sleep | 75.1 (24.3)
  6-Month: Social: number analyzed (Participants) | 168
  6-Month: Social | 89.1 (18.9)
  6-Month: HRQL: number analyzed (Participants) | 168
  6-Month: HRQL | 77.7 (21.2)
  1-Year: Coping: number analyzed (Participants) | 146
  1-Year: Coping | 74.3 (27.5)
  1-Year: Concern: number analyzed (Participants) | 146
  1-Year: Concern | 73.6 (25.6)
  1-Year Sleep: number analyzed (Participants) | 146
  1-Year Sleep | 77.1 (23.0)
  1-Year Social: number analyzed (Participants) | 146
  1-Year Social | 89.0 (18.7)
  1-Year: HRQL: number analyzed (Participants) | 146
  1-Year: HRQL | 77.9 (21.4)

12. Primary Outcome: Performance/Effectiveness - Improvement of Patient UR Symptoms in the Implanted Cohort From Baseline
Description: Change in indication-specific patient symptoms from baseline for all implanted patients by Patient Symptom Questionnaire results. The patient symptoms questionnaire assesses participants' diagnosis-specific symptoms at baseline and at follow-up. Participants who reported a UR diagnosis at baseline were asked about the number of catheterizations required per day.
Time Frame: 6-months, 1-year
Population: Overall number of participants analyzed are those implanted patients who were diagnosed with Urinary Retention (UR). Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: catheterizations per day
Groups:
- Urinary Retention (UR): Patients diagnosed with UR who underwent an Axonics External Trial System (ETS) trial and received an Axonics Implantable Neurostimulator (INS) who experienced fewer catheterizations.
Arm/Group | Urinary Retention (UR)
Number analyzed (Participants) | 50
catheterizations per day
  Baseline: Catheterizations per day | 0.8 (1.8)
  6-month: Catheterizations per day: number analyzed (Participants) | 43
  6-month: Catheterizations per day | 0.2 (0.8)
  1-year: Catheterizations per day: number analyzed (Participants) | 41
  1-year: Catheterizations per day | 0.2 (0.9)

13. Primary Outcome: Performance/Effectiveness - Change in CCF-FIS Score for Participants Diagnosed With FI or With a CCF-FIS Score ≥6 at Baseline
Description: Change in CCF-FIS score at follow-up compared to baseline. Cleveland Clinic Florida - Fecal Incontinence Score (CCF-FIS): includes 5 items (solid, liquid, gas, wears pad and lifestyle alteration) and 5 frequencies (never = 0, rarely = 1, sometimes = 2, usually = 3, always = 4). Scores range from 0 for full continence to 20 for complete incontinence. A higher score indicates more severe FI symptoms and a score ≥ 6 indicates moderate to severe FI symptoms.
Time Frame: 6-months, 1-year
Population: A CCF-FIS was collected for all participants at baseline. At follow-up, a CCF-FIS was only collected for those participants with a FI diagnosis or a CCF-FIS score ≥ 6 at baseline. Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fecal Incontinence (FI): Patients diagnosed with Fecal Incontinence (FI) who were scheduled to undergo an Axonics External Trial System (ETS) trial or receive an Axonics Implantable Neurostimulator (INS)
Arm/Group | Fecal Incontinence (FI)
Number analyzed (Participants) | 81
score on a scale
  Baseline CCF-FIS Score: number analyzed (Participants) | 78
  Baseline CCF-FIS Score | 10.7 (4.1)
  6-Month: CCF-FIS Score: number analyzed (Participants) | 67
  6-Month: CCF-FIS Score | 6.3 (4.5)
  1-Year CCF-FIS Score: number analyzed (Participants) | 52
  1-Year CCF-FIS Score | 6.8 (4.9)

14. Primary Outcome: Performance/Effectiveness - Change in FIQL Score for Participants Diagnosed With FI or With a CCF-FIS Score ≥6 at Baseline in the Implanted Cohort
Description: Change in FIQL score compared to baseline for implanted participants. Fecal Incontinence Quality of Life (FIQL) includes four different subscales: lifestyle, coping/behavior, depression/self-perception and embarrassment. Subscale scores range from 1 to 5, with 1 indicating lower functional status of qualify of life.
Time Frame: 6-months, 1-year
Population: Overall number of participants analyzed are those implanted patients who were diagnosed with Fecal Incontinence (FI) and/or scored >=6 on CCF-FIS. Overall participants analyzed includes those participants that completed the CCF-FIS & FIQL (data point found in Table 9. Assessment Compliance, Week 1-4).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fecal Incontinence (FI): Patients diagnosed with fecal incontinence (FI) who underwent an Axonics External Trial System (ETS) trial and received an Axonics Implantable Neurostimulator (INS) who experienced an increase in scores for all four domains: lifestyle, coping behavior, depression or self-perception, and level of embarrassment.
Arm/Group | Fecal Incontinence (FI)
Number analyzed (Participants) | 81
score on a scale
  Baseline: Lifestyle: number analyzed (Participants) | 75
  Baseline: Lifestyle | 2.7 (1.0)
  Baseline: Coping/Behavior: number analyzed (Participants) | 76
  Baseline: Coping/Behavior | 2.1 (0.8)
  Baseline: Depression/Self Perception: number analyzed (Participants) | 78
  Baseline: Depression/Self Perception | 3.0 (0.9)
  Baseline: Embarrassment: number analyzed (Participants) | 76
  Baseline: Embarrassment | 2.2 (0.9)
  6-Month: Lifestyle: number analyzed (Participants) | 63
  6-Month: Lifestyle | 3.4 (0.8)
  6-Month: Coping/Behavior: number analyzed (Participants) | 62
  6-Month: Coping/Behavior | 2.9 (0.9)
  6-Month: Depression/Self Perception: number analyzed (Participants) | 67
  6-Month: Depression/Self Perception | 3.6 (0.8)
  6-Month: Embarrassment: number analyzed (Participants) | 62
  6-Month: Embarrassment | 3.0 (1.0)
  1-Year: Lifestyle: number analyzed (Participants) | 44
  1-Year: Lifestyle | 3.1 (1.0)
  1-Year: Coping/Behavior: number analyzed (Participants) | 44
  1-Year: Coping/Behavior | 2.7 (0.8)
  1-Year: Depression/Self Perception: number analyzed (Participants) | 51
  1-Year: Depression/Self Perception | 3.7 (0.7)
  1-Year: Embarrassment: number analyzed (Participants) | 45
  1-Year: Embarrassment | 2.7 (1.0)

15. Primary Outcome: Performance/Effectiveness - Changes From Baseline in O'Leary Sant Score for Urinary Frequency Participants in the Implanted Cohort
Description: Change in O'Leary Sant score at follow-up compared to baseline for all implanted participants. The O'Leary Sant is a validated questionnaire designed to provide data on painful bladder and urinary frequency symptoms. Symptom and Problem Index scores are calculated based on responses to two sets of 4 questions with higher scores representing more symptoms/problems. A total score from 0 - 40 is also calculated based on all responses. At follow-up, an O'Leary Sant was only collected for those participants an O'Leary Sant score ≥ 6 at baseline.
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Overactive Bladder (OAB) - Urinary Frequency (UF): Patients diagnosed with overactive bladder (OAB), urinary frequency (UF) who were scheduled to undergo an Axonics External Trial System (ETS) trial or receive an Axonics Implantable Neurostimulator (INS)
Arm/Group | Overactive Bladder (OAB) - Urinary Frequency (UF)
Number analyzed (Participants) | 151
score on a scale
  Baseline: Total Score | 20.7 (6.8)
  6-Month: Total Score | 11.7 (8.2)
  1-Year Total Score: number analyzed (Participants) | 115
  1-Year Total Score | 11.8 (7.7)

16. Primary Outcome: Performance/Effectiveness - Change in AUA-SI Score for Urinary Retention Participants in the Implanted Cohort
Description: Change in AUA-SI score at follow-up compared to baseline for Urinary Retention participants who were implanted with the device. The AUA-SI (American Urological Association Symptom Index) is a questionnaire used to assess the severity of lower urinary tract symptoms (LUTS) in men, with scores ranging from 0 to 35, categorizing symptoms as mild (0-7), moderate (8-19), or severe (20-35). A higher score indicates more severe UR symptoms and a score of greater than 8 indicates moderate to severe UR symptoms.
Time Frame: 6-months, 1-year
Population: Difference in number of participants across timepoints account for study exits that occurred during follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Urinary Retention (UR): Patients diagnosed with urinary retention (UR) who were scheduled to undergo an Axonics External Trial System (ETS) trial or receive an Axonics Implantable Neurostimulator (INS)
Arm/Group | Urinary Retention (UR)
Number analyzed (Participants) | 50
score on a scale
  Baseline: AUA-SI Score | 18.7 (8.6)
  6-Month: AUA-SI Score | 10.4 (8.1)
  1-Year: AUA-SI Score: number analyzed (Participants) | 41
  1-Year: AUA-SI Score | 10.3 (8.4)

17. Primary Outcome: Adverse Event Reporting (Safety)
Description: The number and participant rates of device-related AEs and Serious Adverse Events (SAEs), including Serious Adverse Device Effects (SADEs).
Time Frame: 1-year
Measure: Number; unit: number of events
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
Number analyzed (Participants) | 253
number of events
  Device-related SAEs | 0
  Procedure-related SAEs | 2
  Device- and Procedure-related SAEs | 0
  SAEs (not device- or procedure-related) | 13

ADVERSE EVENTS:
Time Frame: 1 year
Description: This non-randomized study recruited participants who may have had an overlap of their diagnoses, some of which the overlap could have been as a result of their responses to certain questionnaires. For example, participants who scored ≥6 on the CCF-FIS questionnaires at baseline would be included in the FI cohort analysis while their primary indication may be UUI. Because of this, the numbers in the adverse event table are not able to be stratified into each type of diagnosis.
Groups:
- Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI): Patients diagnosed with overactive bladder (OAB), urinary retention (UR), and/or fecal incontinence (FI) who were scheduled to undergo an Axonics External Trial System (ETS) trial or receive an Axonics Implantable Neurostimulator (INS). This non-randomized study recruited participants who may have had an overlap of their diagnoses, some of which the overlap could have been as a result of their responses to certain questionnaires. For example, participants who scored ≥6 on the CCF-FIS questionnaires at baseline would be included in the FI cohort analysis while their primary indication may be UUI. Because of this, the adverse event numbers are not able to be stratified into each type of diagnosis.
Arm/Group | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI)
All-Cause Mortality (participants affected / at risk) | 1/253
Serious Adverse Events (participants affected / at risk) | 14/253
Other Adverse Events (participants affected / at risk) | 20/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI) (N=253)
Transient Ischemic Attack (Nervous system disorders) | 2
Acute Encephalopathy (Nervous system disorders) | 1
Orthostatic Hypotension (Blood and lymphatic system disorders) | 1
Syncope (Nervous system disorders) | 1
Pain at INS Site (Musculoskeletal and connective tissue disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Hypernatremia (Blood and lymphatic system disorders) | 1
Chest Pain (Cardiac disorders) | 1
Exacerbation of Hypokalemic Periodic Paralysis (Musculoskeletal and connective tissue disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Septic Shock (Infections and infestations) | 1
Cerebral Vascular Accident (Nervous system disorders) | 1
Urosepsis (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overactive Bladder (OAB), Urinary Retention (UR), and/or Fecal Incontinence (FI) (N=253)
Uncomfortable/Undesirable Stimulation (Nervous system disorders) | 5
Implant Site Infection (Infections and infestations) | 3
Pain at Lead Site (Skin and subcutaneous tissue disorders) | 2
Pain at INS Site (Skin and subcutaneous tissue disorders) | 2
Implant Site Induration (Skin and subcutaneous tissue disorders) | 1
Lead Erosion (Product Issues) | 1
Lead Migration (Product Issues) | 1
Loss of Efficacy (Nervous system disorders) | 1
Pain at Contralateral Hip (Musculoskeletal and connective tissue disorders) | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 1
Worsening of Chronic Back Pain (Musculoskeletal and connective tissue disorders) | 1
Worsening of Urinary Symptoms (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT05064384/Prot_000.pdf
  • Informed Consent Form (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT05064384/ICF_001.pdf